CLINICAL TRIAL: NCT04076540
Title: A Phase I Randomized, Double-blind Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD4041 Following Single Ascending Dose Administration to Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD4041 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Eolas Therapeutics INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D7460C00001
Record Dates: First submitted 2019-08-06; First posted 2019-09-03 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation
Keywords: Safety; Tolerability; Pharmacokinetics; Healthy Volunteers
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD4041 (Experimental)
  Interventions: Drug: AZD4041
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4041 — Administration by Oral syringe
  Arms: AZD4041
Drug: Placebo — Administration by Oral syringe
  Arms: Placebo

SUMMARY:
This is a Phase I, first-in-human (FIH), single-center, randomized, double-blind, placebo controlled, single ascending dose, sequential group study in healthy vasectomized male and female subjects of non-childbearing potential, aged 18 to 65 years.

ELIGIBILITY:
Inclusion criteria

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form and in this clinical study protocol.
2. Provision of signed and dated, written Informed Consent Form prior to any mandatory study specific procedures, sampling, and analyses.
3. Subjects must be ≥18 and less than or equal to 65 years of age at the time of signing the Informed Consent Form.
4. Individuals who are healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring.
5. Individuals who weigh ≥50 kg and who have a body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
6. Either male or female.
7. Female subjects must have a negative pregnancy test result at screening and check-in and, on admission to the unit, must not be lactating.
8. Female subjects must be of non-childbearing potential, as confirmed at screening by fulfilling one of the following criteria:

   1. Post-menopausal women must have had ≥12 months of spontaneous amenorrhea with a follicle stimulating hormone (FSH) concentration consistently ≥40 mIU/mL and must have a negative pregnancy test result at screening and check-in.
   2. Surgically sterile women, defined as those who have had a hysterectomy, bilateral ovariectomy (oophorectomy), bilateral salpingectomy, or bilateral tubal ligation. Women who are surgically sterile must provide documentation of the procedure by an operative report or relevant medical records, or by ultrasound, and must have a negative pregnancy test result at screening and check-in.
9. Male subjects must be vasectomized.

Exclusion criteria

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History of any significant psychiatric disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (American Psychiatric Association 2013) which, in the opinion of the Investigator, could be detrimental to subject safety or could compromise study data interpretation.
3. Male subjects with a history of oligospermia or azoospermia or any other disorder of the reproductive system.
4. Subjects who are undergoing treatment or evaluation for infertility.
5. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
6. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of administration of Investigational Product.
7. Any clinically important abnormalities noted at the screening assessments in clinical chemistry, hematology, or urinalysis results as judged by the Investigator.
8. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus antibodies.
9. Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

   1. Systolic BP <90 mmHg or ≥140 mmHg.
   2. Diastolic BP <50 mmHg or ≥90 mmHg.
   3. HR <45 or >85 beats per minute.
10. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG which, in the Investigator's opinion, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology.
11. ECG interval measured from the onset of the QRS complex to the end of the T wave (QT) interval corrected for HR using Fridericia's formula (QTcF) >450 ms or family history of long QT syndrome.
12. ECG interval measured from the onset of the P wave to the onset of the QRS complex (PR[PQ]) interval shortening <120 ms (PR >110 ms but <120 ms is acceptable if there is no evidence of ventricular pre-excitation).
13. PR(PQ) interval prolongation (>240 ms), persistent or intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.
14. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with ECG interval measured from the onset of the QRS complex to the J point (QRS) >110 ms. Subjects with QRS >110 ms but <115 ms are acceptable if there is no evidence of, eg, ventricular hypertrophy or pre-excitation.
15. Known or suspected history of drug abuse as judged by the Investigator.
16. Current smokers or those who have smoked or used nicotine products within the previous 3 months.
17. History of alcohol abuse or excessive intake of alcohol defined as an average weekly intake of >21 units or an average daily intake of >3 units for men or an average weekly intake of >14 units or an average daily intake of >2 units for women. One unit is equivalent to a half pint (250 mL) of beer, 1 measure (25 mL) of spirits, or 1 glass (125 mL) of wine. If a subject is currently diagnosed with abuse of or dependence on alcohol, the subject will not be allowed to enroll in the study, unless the alcohol abuse/dependence is in full (complete, not partial), sustained (>1 year) remission.
18. Positive screen for drugs of abuse at screening or admission to the unit or positive screen for alcohol at screening to the unit prior to administration of IP.
19. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4041.
20. Plasma donation within 1 month of screening or any blood donation/blood loss >500 mL during the 3 months prior to screening.
21. Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the Investigator.
22. Use of drugs with enzyme inducing properties, such as St John's wort, within 3 weeks prior to administration of IP.
23. Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to administration of IP or longer if the medication has a long half life.
24. Use of any prescribed or nonprescribed oral and topical inhibitors/inducers of CYP3A4 (including shampoo).
25. Use of hormone replacement therapy.
26. Subjects who have previously received AZD4041.
27. Has received another new chemical entity (defined as a compound that has not been approved for marketing) within 3 months of administration of IP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit, whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous Phase I study, are not excluded.
28. Involvement of any AstraZeneca or study site employee or their close relatives.
29. Judgement by the Investigator that the subject should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
30. Subjects who are vegans or have medical dietary restrictions.
31. Subjects who cannot communicate reliably with the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca N. Wood-Horrall, MD, Principal Investigator — PPD Development, LP; Darin Brimhall, DO, FACP, Principal Investigator — PPD Development, LP
Locations (2):
- United States (2):
  - Research Site, Las Vegas, Nevada
  - Research Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymised individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de- identified individual patient-level data in an approved sponsor tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7460C00001&attachmentIdentifier=5c22ca47-e770-4094-a6d7-3722b140f995&fileName=D7460C00001_CSR_Synopsis_Redacted_PDF-A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Pooled Placebo: Single dose oral solution pooled from 6 cohorts
- AZD4041 X mg; AZD4041 3X mg; AZD4041 9X mg; AZD4041 20X mg; AZD4041 40X mg; AZD4041 80X mg: Single dose oral solution
Period: Cohort 1: Dose Level X
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Started (8) | 2 | 6 | 0 | 0 | 0 | 0 | 0
Completed (8) | 2 | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: Dose Level 3X
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Started (8) | 2 | 0 | 6 | 0 | 0 | 0 | 0
Completed (8) | 2 | 0 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3: Dose Level 9X
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Started (8) | 2 | 0 | 0 | 6 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 4: Dose Level 20X
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Started (8) | 2 | 0 | 0 | 0 | 6 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 5: Dose Level 40X
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Started | 2 | 0 | 0 | 0 | 0 | 6 | 0
Completed | 2 | 0 | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 6: Dose Level 80X
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Started | 2 | 0 | 0 | 0 | 0 | 0 | 6
Completed | 2 | 0 | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (12.26) | 49.8 (11.81) | 37.3 (14.49) | 46.0 (14.99) | 55.5 (4.85) | 46.2 (8.68) | 53.5 (11.67) | 47.7 (50.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 1 | 2 | 5 | 4 | 5 | 25
  Male | 7 | 3 | 5 | 4 | 1 | 2 | 1 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 3 | 1 | 2 | 3 | 17
  Not Hispanic or Latino | 9 | 3 | 4 | 3 | 5 | 4 | 3 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 1 | 1 | 1 | 1 | 1 | 11
  White | 7 | 5 | 4 | 5 | 3 | 5 | 5 | 34
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 75.45 (10.62) | 75.23 (13.923) | 69.47 (9.92) | 74.37 (14.05) | 67.62 (15.47) | 78.58 (8.63) | 61.03 (10.28) | 72.15 (12.34)
Height [Mean (Standard Deviation); unit: cm] | 169.96 (9.37) | 166.13 (12.51) | 167.70 (8.31) | 165.17 (9.55) | 164.88 (9.160) | 174.40 (6.53) | 159.02 (9.42) | 167.15 (9.78)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.14 (3.11) | 27.02 (1.87) | 24.63 (2.60) | 27.07 (2.72) | 24.68 (3.84) | 25.85 (2.50) | 24.00 (2.03) | 25.69 (2.82)

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Number of participants experiencing any adverse event
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 5 | 0 | 1 | 1 | 1 | 3 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Number of participants experiencing any treatment emergent adverse events
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 5 | 0 | 1 | 1 | 1 | 3 | 1

3. Primary Outcome: Number of Participants With Treatment-Related TEAEs
Description: Number of participants experiencing any treatment-related TEAEs
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 1 | 0 | 1 | 1 | 0 | 2 | 0

4. Primary Outcome: Number of Participants With Moderate TEAEs
Description: Number of participants experiencing any moderate TEAEs
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 1 | 0 | 0 | 2 | 0

5. Primary Outcome: Number of Participants With Treatment-Related Moderate TEAEs
Description: Number of participants experiencing any treatment-related moderate TEAEs
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 1 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Severe TEAEs
Description: Number of participants experiencing any severe TEAEs
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Treatment-Related Severe TEAEs
Description: Number of participants experiencing any treatment-related severe TEAEs
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants experiencing any serious adverse events (SAEs)
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Treatment-Related SAEs
Description: Number of participants experiencing any treatment-related serious adverse events (SAEs)
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With TEAEs Leading to Early Discontinuation
Description: Number of participants with treatment-emergent adverse events leading to early discontinuation
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participant Deaths
Description: Number of participants who died
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Abnormal Vital Signs
Description: Number of participants with treatment-related abnormal vital signs considered clinically significant or reported as a treatment-emergent adverse event by the investigator.
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 2 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Abnormal Vital Signs (Blood Pressure)
Description: Number of participants with treatment-related abnormal blood pressure considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Abnormal Vital Signs (Heart Rate)
Description: Number of participants with treatment-related abnormal heart rate considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Pulse Rate at Baseline and Day 1 2 Hours Post.
Description: Measured by standing pulse rate at baseline and 2 hours post
Time Frame: Baseline and Day 1
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Beats per minute
  Baseline | 77.8 (9.53) | 74.8 (8.45) | 82.2 (9.77) | 90.7 (7.34) | 83.5 (10.01) | 78.2 (9.43) | 82.3 (23.95)
  Day 1 (2 hours) | 81.7 (14.18) | 80.2 (8.04) | 83.7 (10.13) | 102.8 (31.16) | 78.2 (10.05) | 82.0 (18.31) | 90.3 (15.71)

16. Primary Outcome: Number of Participants With Abnormal Safety Laboratory Tests (Hematology)
Description: Number of participants with treatment-related abnormal hematology values considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Abnormal Safety Laboratory Tests (Serum Chemistry)
Description: Number of participants with treatment-related abnormal serum chemistry values considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Abnormal Safety Laboratory Tests (Urinalysis)
Description: Number of participants with treatment-related abnormal urinalysis values considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: 6 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Cmax of AZD4041
Description: Maximum (peak) plasma concentration of AZD4041
Time Frame: Thru Day 4
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 14.7 (15.0) | 44.6 (37.9) | 154 (24.7) | 382 (21.2) | 620 (25.9) | 1060 (26.0)

20. Primary Outcome: Number of Participants With Abnormal 12-lead ECGs
Description: Number of participants with abnormal 12-lead electrocardiograms (ECGs), considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: 4 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 1 | 0

21. Primary Outcome: Heart Rate at Baseline and Times Post Dose
Description: Measured by digital electrocardiograms (ECGs)
Time Frame: Thru Day 4
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Beats per minute
  Baseline | 60.7 (6.5) | 63.0 (4.0) | 53.7 (5.4) | 67.3 (5.7) | 64.2 (4.9) | 66.0 (6.3) | 61.7 (8.21)
  Day 1 (0.5 hour) | 58.6 (4.7) | 64.0 (4.3) | 55.8 (5.0) | 67.8 (8.9) | 65.3 (6.7) | 61.2 (6.4) | 57.7 (8.24)
  Day 1 (1 hour) | 59.0 (5.0) | 62.5 (5.8) | 56.2 (5.0) | 67.0 (8.7) | 62.7 (5.2) | 60.8 (8.0) | 67.5 (7.4)
  Day 1 (1.5 hours) | 58.3 (5.8) | 62.5 (5.6) | 56.0 (4.2) | 66.0 (9.0) | 62.8 (5.9) | 61.7 (8.4) | 57.8 (11.2)
  Day 1 (2 hours) | 57.8 (4.8) | 63.2 (6.8) | 55.8 (7.4) | 67.2 (8.8) | 61.7 (5.9) | 61.0 (8.3) | 57.8 (8.30)
  Day 1 (3 hours) | 58.0 (5.6) | 65.5 (6.8) | 56.7 (5.16) | 67.0 (7.4) | 62.3 (5.1) | 63.2 (7.0) | 58.3 (9.0)
  Day 1 (4 hours) | 68.7 (5.9) | 64.7 (7.2) | 56.5 (4.1) | 66.2 (7.9) | 64.0 (5.1) | 61.0 (8.1) | 57.3 (7.8)
  Day 1 (6 hours) | 67.1 (6.02) | 72.7 (7.26) | 63.0 (6.23) | 76.3 (6.06) | 73.8 (7.91) | 65.7 (8.45) | 62.0 (11.51)
  Day 1 (8 hours) | 63.5 (6.8) | 68.7 (5.2) | 59.7 (6.2) | 73.5 (12.1) | 67.7 (7.2) | 64.0 (9.0) | 62.3 (11.2)
  Day 1 (12 hours) | 63.8 (6.8) | 66.5 (6.3) | 61.7 (8.3) | 74.8 (9.9) | 73.2 (6.6) | 65.7 (10.2) | 60.7 (10.0)
  Day 2 (24 hours) | 61.8 (6.9) | 66.2 (6.2) | 57.2 (7.2) | 68.0 (8.3) | 68.3 (7.1) | 62.5 (8.5) | 61.3 (8.5)
  Day 2 (36 hours) | 65.0 (7.2) | 65.5 (8.3) | 61.2 (4.6) | 71.0 (9.6) | 73.0 (10.1) | 67.8 (8.9) | 61.0 (9.6)
  Day 3 (48 hours) | 62.8 (5.64) | 67.3 (7.87) | 57.7 (3.20) | 68.8 (7.22) | 66.7 (6.89) | 65.7 (8.80) | 62.2 (12.73)
  Day 4 (Day 4 analysis only applicable for arms C,D and E) | 62.8 (9.9) | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and Erts. | 69.0 (9.21) | 66.0 (6.66) | 61.3 (7.55)

22. Primary Outcome: Aggregate P-R Interval at Baseline and Time Post Dose
Description: PR interval is the time from the beginning of atrial depolarization to the onset of ventricular depolarization. Measured by digital electrocardiograms (ECGs)
Time Frame: Thru Day 4
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
milliseconds
  Baseline | 152.1 (8.16) | 150.5 (7.06) | 170.8 (14.47) | 154.0 (18.90) | 153.5 (19.73) | 153.8 (7.81) | 154.5 (27.05)
  Day 1 (0.5 hour) | 152.3 (9.18) | 148.5 (7.53) | 169.2 (12.77) | 158.5 (20.63) | 152.0 (17.18) | 156.0 (11.03) | 156.3 (26.88)
  Day 1 (1 hour) | 151.9 (7.66) | 151.5 (9.16) | 170.3 (12.37) | 157.0 (21.82) | 151.7 (16.97) | 159.7 (12.91) | 158.7 (25.63)
  Day 1 (1.5 hours) | 150.9 (7.54) | 151.0 (8.97) | 169.2 (12.27) | 158.8 (21.66) | 151.0 (16.76) | 159.2 (11.30) | 158.5 (25.27)
  Day 1 (2 hours) | 151.8 (8.67) | 151.2 (9.00) | 170.8 (12.75) | 159.5 (21.06) | 151.2 (17.02) | 160.5 (12.18) | 156.8 (25.87)
  Day 1 (3 hours) | 153.7 (9.78) | 151.3 (7.42) | 166.2 (10.93) | 158.5 (22.06) | 150.8 (15.99) | 156.3 (14.71) | 158.7 (28.68)
  Day 1 (4 hours) | 151.6 (8.02) | 151.2 (9.56) | 165.0 (10.49) | 157.5 (24.83) | 150.3 (15.56) | 159.8 (10.46) | 159.0 (28.47)
  Day 1 (6 hours) | 150.4 (8.75) | 145.5 (8.83) | 160.7 (7.23) | 152.7 (19.75) | 144.2 (12.77) | 155.0 (9.12) | 154.7 (20.27)
  Day 1 (8 hours) | 150.7 (7.98) | 146.5 (7.97) | 162.8 (8.93) | 155.0 (20.01) | 146.8 (13.64) | 155.7 (9.75) | 153.3 (23.76)
  Day 1 (12 hours) | 150.1 (6.97) | 151.5 (6.35) | 163.7 (9.37) | 156.0 (19.27) | 147.8 (12.77) | 160.2 (12.88) | 155.8 (25.35)
  Day 2 (24 hours) | 148.7 (5.52) | 151.5 (8.67) | 166.5 (15.40) | 156.3 (19.50) | 151.3 (18.78) | 155.8 (10.23) | 155.5 (14.21)
  Day 2 (36 hours) | 151.9 (6.14) | 152.8 (9.35) | 163.5 (12.01) | 161.7 (20.10) | 151.3 (17.96) | 156.0 (8.10) | 158.3 (26.52)
  Day 3 (48 hours) | 150.8 (9.30) | 149.7 (6.44) | 170.3 (12.44) | 157.2 (19.91) | 152.3 (17.28) | 156.3 (11.54) | 161.0 (28.62)
  Day 4 (Day 4 analysis only applicable for arms C,D and E) | 150.8 (10.5) | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | 156.3 (19.67) | 155.3 (11.38) | 160.2 (25.23)

23. Primary Outcome: Aggregate QRS Complex at Baseline and Times Post Dose
Description: QRS complex represents the electrical impulse as it spreads through the ventricles and indicates ventricular depolarization. Measured by digital electrocardiograms (ECGs)
Time Frame: Thru Day 4
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
milliseconds
  Baseline | 91.1 (8.67) | 89.5 (9.33) | 95.3 (8.82) | 90.2 (7.57) | 87.7 (6.02) | 87.7 (8.50) | 88.0 (9.53)
  Day 1 (0.5 hour) | 90.5 (9.66) | 89.3 (8.94) | 94.5 (8.34) | 89.8 (8.11) | 87.7 (6.28) | 88.0 (10.49) | 88.5 (9.27)
  Day 1 (1 hour) | 91.7 (9.40) | 90.9 (8.41) | 94.3 (8.52) | 91.3 (9.44) | 88.5 (6.09) | 87.5 (8.92) | 87.7 (9.24)
  Day 1 (1.5 hours) | 90.7 (9.25) | 90.3 (8.82) | 93.8 (8.89) | 90.7 (8.66) | 87.5 (7.37) | 87.8 (10.42) | 88.5 (8.76)
  Day 1 (2 hours) | 91.3 (9.18) | 89.7 (8.73) | 93.7 (9.73) | 89.5 (8.62) | 88.5 (6.02) | 88.0 (9.67) | 88.7 (8.50)
  Day 1 (3 hours) | 91.0 (9.80) | 89.8 (8.66) | 94.0 (8.37) | 90.3 (7.79) | 88.0 (7.46) | 88.0 (11.30) | 89.5 (8.92)
  Day 1 (4 hours) | 91.1 (9.54) | 89.7 (8.31) | 93.5 (8.09) | 91.0 (9.08) | 88.3 (6.62) | 88.5 (10.41) | 89.2 (7.83)
  Day 1 (6 hours) | 90.3 (8.97) | 89.3 (8.07) | 92.0 (10.18) | 90.5 (10.01) | 84.8 (7.47) | 88.3 (11.25) | 85.0 (10.04)
  Day 1 (8 hours) | 90.3 (9.00) | 88.7 (9.20) | 92.0 (9.72) | 89.3 (9.85) | 86.7 (7.03) | 87.7 (11.62) | 87.7 (8.52)
  Day 1 (12 hours) | 90.8 (9.30) | 89.7 (8.96) | 92.2 (10.78) | 89.8 (9.83) | 87.2 (8.26) | 89.2 (9.93) | 89.8 (8.93)
  Day 2 (24 hours) | 90.4 (8.53) | 88.7 (7.34) | 94.0 (8.60) | 89.8 (8.73) | 85.7 (6.56) | 87.8 (9.50) | 86.5 (9.54)
  Day 2 (36 hours) | 90.2 (10.08) | 89.8 (8.98) | 91.5 (8.98) | 91.3 (9.18) | 87.2 (8.13) | 37.7 (7.74) | 80.0 (8.12)
  Day 3 (48 hours) | 88.6 (8.99) | 88.0 (8.46) | 93.2 (8.42) | 90.2 (8.38) | 86.8 (7.17) | 86.0 (7.87) | 89.7 (8.50)
  Day 4 (Day 4 analysis only applicable for arms C,D and E) | 35.7 (6.38) | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | 87.3 (7.79) | 86.8 (8.52) | 89.8 (7.60)

24. Primary Outcome: Aggregate QT Interval at Baseline and Times Post Dose
Description: The QT interval is measured from the beginning of the QRS complex to the end of the T wave and primarily represents the return of stimulated ventricles to their resting state (ventricular repolarization). Measured by digital electrocardiograms (ECGs)
Time Frame: Thru Day 4
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
milliseconds
  Baseline | 382.5 (29.29) | 377.8 (21.61) | 389.5 (27.27) | 359.2 (13.50) | 366.3 (17.66) | 389.2 (10.21) | 402.2 (29.91)
  Day 1 (0.5 hour) | 384.5 (31.22) | 374.8 (18.88) | 379.8 (22.42) | 357.0 (13.89) | 363.0 (11.76) | 396.3 (7.26) | 405.3 (30.58)
  Day 1 (1 hour) | 389.9 (31.50) | 380.8 (19.08) | 381.5 (24.83) | 362.5 (16.63) | 373.2 (16.09) | 404.3 (7.23) | 410.5 (30.07)
  Day 1 (1.5 hours) | 390.0 (30.11) | 388.7 (19.94) | 382.5 (24.70) | 364.2 (15.77) | 374.5 (12.77) | 406.5 (15.90) | 413.8 (34.60)
  Day 1 (2 hours) | 391.8 (28.72) | 383.5 (20.52) | 383.8 (25.19) | 362.3 (17.60) | 377.2 (14.55) | 411.0 (9.36) | 417.0 (31.28)
  Day 1 (3 hours) | 390.6 (30.40) | 382.0 (21.14) | 380.3 (18.36) | 363.2 (13.32) | 376.7 (16.60) | 405.8 (12.50) | 413.0 (31.93)
  Day 1 (4 hours) | 391.8 (30.12) | 384.8 (17.95) | 381.2 (21.98) | 367.7 (16.17) | 374.3 (21.40) | 408.3 (11.86) | 415.8 (32.68)
  Day 1 (6 hours) | 369.3 (24.74) | 356.5 (21.50) | 364.2 (17.93) | 346.0 (13.25) | 345.0 (21.95) | 386.2 (13.23) | 387.0 (29.05)
  Day 1 (8 hours) | 377.9 (26.52) | 363.0 (12.43) | 371.0 (26.60) | 349.0 (14.60) | 359.7 (20.20) | 391.0 (15.94) | 391.8 (36.66)
  Day 1 (12 hours) | 377.7 (27.94) | 371.7 (13.85) | 367.8 (29.36) | 350.3 (10.41) | 356.5 (23.67) | 389.7 (13.22) | 399.8 (34.52)
  Day 2 (24 hours) | 380.4 (22.44) | 370.2 (20.31) | 374.3 (24.06) | 359.0 (15.74) | 358.0 (19.71) | 396.2 (20.59) | 400.8 (27.33)
  Day 2 (36 hours) | 375.2 (28.50) | 373.2 (13.42) | 363.8 (15.88) | 358.5 (13.28) | 357.0 (21.25) | 390.8 (20.13) | 399.2 (30.42)
  Day 3 (48 hours) | 377.8 (23.95) | 266.0 (19.05) | 274.8 (21.45) | 357.8 (16.20) | 366.3 (17.81) | 391.7 (16.77) | 402.7 (36.53)
  Day 4 (Day 4 analysis only applicable for arms C,D and E) | 379.5 (40.02) | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | 357.8 (21.15) | 392.2 (23.99) | 404.7 (30.59)

25. Primary Outcome: Aggregate QTcF Interval and Times Post Dose
Description: The QTcF if the QT interval corrected for heart rate using Fridercia's formula. Measured by digital electrocardiograms (ECGs)
Time Frame: Thru Day 4
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
milliseconds
  Baseline | 382.9 (23.45) | 383.3 (20.29) | 374.8 (23.63) | 372.8 (15.41) | 374.7 (21.39) | 402.0 (17.34) | 404.7 (18.98)
  Day 1 (0.5 hour) | 381.0 (38.33) | 382.7 (18.5) | 370.0 (21.96) | 371.0 (17.85) | 373.2 (20.37) | 398.7 (14.50) | 398.0 (17.79)
  Day 1 (1 hour) | 387.0 (38.04) | 385.3 (20.61) | 372.7 (23.57) | 375.0 (19.31) | 378.7 (20.78) | 405.3 (18.95) | 403.3 (22.06)
  Day 1 (1.5 hours) | 385.9 (26.62) | 393.7 (23.39) | 374.0 (25.20) | 375.2 (18.32) | 380.5 (20.32) | 409.3 (20.03) | 405.8 (19.46)
  Day 1 (2 hours) | 386.6 (25.90) | 389.8 (22.93) | 374.0 (26.27) | 375.7 (18.48) | 380.0 (21.35) | 411.7 (18.08) | 409.7 (22.05)
  Day 1 (3 hours) | 385.6 (26.61) | 392.8 (23.78) | 373.0 (23.44) | 376.3 (18.45) | 381.5 (21.78) | 411.8 (16.80) | 407.2 (19.65)
  Day 1 (4 hours) | 388.0 (24.80) | 394.2 (23.27) | 373.2 (23.02) | 379.5 (17.21) | 382.3 (19.76) | 409.7 (16.78) | 407.8 (21.86)
  Day 1 (6 hours) | 382.8 (20.70) | 379.3 (21.29) | 369.7 (17.74) | 374.7 (16.39) | 369.0 (17.73) | 396.7 (13.47) | 388.8 (13.82)
  Day 1 (8 hours) | 383.9 (20.34) | 380.0 (17.52) | 369.8 (22.20) | 371.8 (15.25) | 373.7 (16.23) | 398.5 (19.93) | 393.7 (16.23)
  Day 1 (12 hours) | 384.5 (23.77) | 384.2 (14.47) | 369.7 (23.24) | 376.2 (12.83) | 380.0 (20.31) | 400.5 (9.59) | 399.0 (17.05)
  Day 2 (24 hours) | 382.2 (21.46) | 381.7 (20.07) | 367.3 (20.22) | 373.8 (18.37) | 373.3 (19.73) | 400.8 (19.16) | 402.3 (20.56)
  Day 2 (36 hours) | 384.3 (21.21) | 383.3 (17.85) | 366.0 (14.38) | 378.3 (14.32) | 379.8 (17.62) | 406.3 (22.34) | 399.2 (9.72)
  Day 3 (48 hours) | 383.0 (20.91) | 379.5 (17.21) | 269.3 (18.54) | 373.8 (16.39) | 379.0 (18.87) | 402.7 (17.39) | 404.3 (13.65)
  Day 4 (Day 4 analysis only applicable for arms C,D and E) | 383.0 (27.25) | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E cohorts | 374.2 (16.77) | 403.8 (20.09) | 406.0 (17.60)

26. Primary Outcome: Aggregate RR Interval at Baseline and Times Post Dose
Description: The RR interval the time elapsed between two successive R waves of the QRS signal on the electrocardiogram. Measured by digital electrocardiograms (ECGs)
Time Frame: Thru Day 4
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
milliseconds
  Baseline | 998.9 (94.86) | 957.5 (55.03) | 1126.0 (123.29) | 896.5 (76.66) | 939.0 (70.03) | 913.0 (85.26) | 985.0 (127.74)
  Day 1 (0.5 hour) | 1029.6 (78.39) | 942.0 (62.03) | 1086.3 (105.03) | 898.7 (124.48) | 927.0 (90.52) | 988.2 (111.95) | 1059.8 (153.49)
  Day 1 (1 hour) | 1023.9 (81.90) | 968.3 (89.63) | 1075.8 (105.83) | 912.0 (132.25) | 962.0 (74.11) | 1003.5 (139.04) | 1057.8 (138.05)
  Day 1 (1.5 hours) | 1035.2 (95.40) | 965.5 (84.72) | 1074.2 (95.98) | 922.3 (134.42) | 960.7 (89.40) | 989.7 (144.62) | 1071.5 (207.00)
  Day 1 (2 hours) | 1043.1 (81.48) | 958.0 (107.71) | 1089.3 (148.54) | 904.7 (121.65) | 983.3 (99.76) | 1003.5 (141.24) | 1059.3 (152.01)
  Day 1 (3 hours) | 1041.4 (100.88) | 925.2 (94.41) | 1066.3 (96.37) | 905.0 (101.31) | 966.5 (85.55) | 965.2 (123.68) | 1048.8 (158.48)
  Day 1 (4 hours) | 1030.5 (101.07) | 938.3 (102.44) | 1068.2 (78.58) | 916.2 (112.82) | 941.8 (71.97) | 998.7 (145.89) | 1063.7 (145.71)
  Day 1 (6 hours) | 900.5 (80.31) | 832.7 (83.65) | 959.5 (74.07) | 790.0 (63.33) | 819.2 (86.55) | 929.7 (128.82) | 996.2 (184.44)
  Day 1 (8 hours) | 955.1 (100.17) | 875.8 (67.69) | 1012.3 (101.19) | 837.0 (147.36) | 894.8 (92.50) | 955.0 (139.11) | 990.5 (178.05)
  Day 1 (12 hours) | 950.9 (102.54) | 909.2 (85.41) | 899.0 (129.62) | 813.8 (144.25) | 826.3 (76.49) | 929.8 (147.80) | 1012.3 (172.32)
  Day 2 (24 hours) | 990.7 (112.51) | 915.3 (90.73) | 1064.0 (139.41) | 891.3 (103.62) | 884.7 (94.73) | 973.8 (139.99) | 994.7 (141.06)
  Day 2 (36 hours) | 931.5 (102.06) | 930.3 (130.67) | 985.0 (78.92) | 856.7 (111.45) | 836.0 (110.22) | 897.8 (125.72) | 1004.0 (170.62)
  Day 3 (48 hours) | 960.9 (81.90) | 900.3 (101.70) | 1044.5 (57.48) | 881.5 (95.33) | 906.8 (88.49) | 928.2 (134.76) | 996.0 (196.50)
  Day 4 (Day 4 analysis only applicable for arms C,D and E) | 973.3 (142.46) | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | NA (NA) — Day 4 analysis only applicable for arms C,D and E | 879.0 (106.47) | 918.3 (94.50) | 991.7 (118.28)

27. Primary Outcome: Number of Participants With Abnormal Testosterone Test Results
Description: Number of participants with abnormal testosterone levels test results, considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: Thru Day 4
Population: Safety Analysis Set (Performed only in males recruited after protocol amendment)
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 1 | 1 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

28. Primary Outcome: Number of Participants With Abnormal Luteinizing Hormone Test Results
Description: Number of participants with abnormal luteinizing hormone (LH) levels test results, considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: Thru Day 4
Population: Safety Analysis Set (Performed only in males recruited after protocol amendment)
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 1 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Primary Outcome: Number of Participants With Abnormal Follicle Stimulating Hormone Test Results
Description: Number of participants with abnormal follicle stimulating hormone (FSH) levels test results, considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: Thru Day 4
Population: Safety Analysis Set (Performed only in males recruited after protocol amendment)
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 1 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Primary Outcome: Number of Participants With Abnormal Inhibin B Test Results
Description: Number of participants with abnormal Inhibin B levels test results, considered clinically significant or reported as a treatment-emergent adverse event by the investigator
Time Frame: Thru Day 4
Population: Safety Analysis Set (Performed only in males recruited after protocol amendment)
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 1 | 1 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Tmax of AZD4041
Description: Time to reach maximum (peak) plasma concentration of AZD4041
Time Frame: Thru Day 4
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour
Arm/Group | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour | 0.50 [0.50 to 1.00] | 1.00 [0.50 to 2.02] | 0.50 [0.50 to 0.50] | 1.00 [0.50 to 1.15] | 1.00 [0.25 to 1.55] | 1.00 [0.50 to 2.00]

32. Secondary Outcome: AUC0-t
Description: Area under the curve of AZD4041 from time 0 to time t (AUC from zero to the last measurable concentration)
Time Frame: Thru Day 4
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hour/mL
Arm/Group | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng·hour/mL | 158 (22.8) | 585 (49.1) | 1790 (29.4) | 5510 (45.6) | 8460 (34.8) | 14400 (27.4)

33. Secondary Outcome: AUC0-inf
Description: Extrapolation of the area under the curve of AZD4041 from zero to infinity
Time Frame: Thru Day 4
Population: Pharmacokinetic Analysis Set. Note AUC0-inf values were excluded where AUCExtrap was >20%
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hour/mL
Arm/Group | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 3 | 5 | 3 | 6 | 6 | 5
ng·hour/mL | 192 (14.7) | 539 (35.8) | 1660 (38.9) | 5950 (52.4) | 9270 (41.0) | 14800 (31.6)

34. Secondary Outcome: t1/2λz
Description: Terminal half-life of AZD4041
Time Frame: Thru Day 4
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
hour | 17.9 (19.0) | 13.0 (40.5) | 19.9 (44.7) | 17.9 (37.9) | 19.8 (33.3) | 16.0 (22.8)

35. Secondary Outcome: CL/F (Volume/Time)
Description: Apparent total clearance of the AZD4041 from plasma
Time Frame: Thru Day 4
Population: Pharmacokinetic Analysis Set. Note CL/V values were excluded where AUCExtrap was >20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 3 | 5 | 3 | 6 | 6 | 5
L/hour | 2.6 (14.7) | 2.8 (35.8) | 2.7 (38.9) | 1.68 (52.4) | 2.16 (41.0) | 2.70 (31.6)

36. Secondary Outcome: Vss/F (Plasma)
Description: Apparent volume of distribution of AZD4041 at steady state
Time Frame: Thru Day 4
Population: Pharmacokinetic Analysis Set. Note Vss/F values were excluded where AUCExtrap was >20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
Number analyzed (Participants) | 3 | 5 | 3 | 6 | 6 | 5
L | 68.8 (4.2) | 45.4 (26.2) | 56.0 (22.9) | 43.3 (22.1) | 61.7 (22.1) | 57.2 (24.3)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Pooled Placebo | AZD4041 X mg | AZD4041 3X mg | AZD4041 9X mg | AZD4041 20X mg | AZD4041 40X mg | AZD4041 80X mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/12 | 0/6 | 1/6 | 1/6 | 1/6 | 3/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=12) | AZD4041 X mg (N=6) | AZD4041 3X mg (N=6) | AZD4041 9X mg (N=6) | AZD4041 20X mg (N=6) | AZD4041 40X mg (N=6) | AZD4041 80X mg (N=6)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Three participants (1 participant in AZD4041 20X mg and 2 participants in AZD4041 40X mg) had 7 important protocol deviations during the study under the category of study procedure and assessments. None were determined by the investigator and sponsor to affect participant safety or the analyses and outcomes of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT04076540/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT04076540/SAP_001.pdf